CLINICAL TRIAL: NCT00472602
Title: Pathogenesis of Liver Fluke Induced Cancer in Thailand
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0001
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2014-07

CONDITIONS: Opisthorchis Viverrini
Keywords: Opisthorchis viverrini, liver fluke, Thailand, cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Opisthorchis viverrini (OV) is a parasite that individuals get from eating raw fish. Infections with this parasite have been associated with liver abnormalities that sometimes lead to bile duct cancer. The purpose of this study is to find out how many people in several areas of the Khon Kaen province are infected with OV, what affect this parasite has on the liver, how the immune system reacts to infection with this parasite, and how the liver is 12 months after being treated for this parasite. Study participants will include 6,000 volunteers, ages 20-60, living in villages surrounding Khon Kaen that have large numbers of people infected with OV. Study procedures will include a stool sample, an ultrasound (sound waves bounced off internal organs to create a picture), and a blood sample. Individuals found to test positive for the parasite will be treated at their local primary health care unit. Participants will be involved in study procedures for up to 12 months.

DETAILED DESCRIPTION:
Liver fluke infection caused by Opisthorchis viverrini (OV) is a major public health problem in parts of East Asia. In Thailand, an estimated 6 million are people infected with OV. Experimental and epidemiological evidence strongly implicate OV infection in the etiology of cholangiocarcinoma (CCA). Studies have shown 10-20% of OV-infected persons have advanced periportal fibrosis (HBA) that progresses to CCA. OV infection may cause inflammation of the bile ducts that results in DNA damage of the epithelium and subsequent malignant transformation. The primary objective of this study is to determine if in-vitro levels of inflammatory cytokines induced by crude antigen extracts of OV are associated with the hepatobiliary abnormalities known to progress to CCA in OV-infected adults aged 20 to 60 years of age. The secondary objective is to determine if in-vitro levels of inflammatory cytokines induced by crude antigen extracts of OV in adults with hepatobiliary abnormalities change 12 months after treatment with praziquantel and if these changes are associated with persistent advanced fibrosis (grade 2 or 3) as determined by ultrasonography. The primary outcome measure is elevated levels of inflammatory cytokines (such as TNF-alpha) induced by OV infection are associated with a 50% greater risk (OR = 1.50) of having advanced fibrosis (grade 2 or 3) as determined by ultrasonography. The secondary outcome measure is elevated levels of inflammatory cytokines 12 months after treatment for OV infection are associated with a 50% greater risk (OR = 1.50) of maintaining the advanced fibrosis that is known to progress to CCA over this time period. District health outposts reporting greater than or equal to 20 percent prevalence of OV infection among adults will be identified, whereupon males and females, 20 to 60 years of age, will be screened for OV infection. Study sites in Thailand will be districts of Ban Pai, Chonnabot, Muncha Khiri and Kok Pochai, regions along the drainage of the Chi River, in the vicinity of the regional capitol, Khon Kaen city. A recruitment ceiling of 20,000 individuals will be established to screen for infection with OV, with 6,000 enrolled in the observational and longitudinal parts of the study. OV-infected individuals will receive an ultrasound examination that will be graded as either HBA positive (advanced fibrosis) or HBA negative (non-advanced fibrosis). Over a 24 month period, 1,116 OV-infected individuals who are HBA positive will be recruited. The first 484 OV-infected individuals with HBA will be age and sex matched with OV-infected individuals from the same region who are HBA negative. Blood samples will be drawn from all volunteers and used in immunological evaluations of OV infection in relation to HBA status. This will constitute the observation stage of the study. The 1,116 OV-infected individuals with HBA will be followed for an additional 12 months, with an ultrasound exam and a blood draw. This will constitute the longitudinal stage of the study. All volunteers will then be treated for OV infection with praziquantel.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 20 and 60 years of age, inclusive, infected with Opisthorchis viverrini
2. Willingness to participate in the study as evidenced by signing the informed consent document.

Exclusion Criteria:

1. Inability to correctly answer all questions on the informed consent comprehension questionnaire.
2. Attends school or works full-time outside of the study area.
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.
4. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer to participate in the trial or would render the subject unable to comply with the protocol.
5. A positive urine Beta-hCG pregnancy test for females.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 695 (Actual)
Dates: Start 2007-08-06; Primary Completion 2012-04-30 (Actual); Study Completion 2012-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand